CLINICAL TRIAL: NCT03918083
Title: WILD (WILD = Wellness Interventions for Life's Demands) 5 Wellness: A 30-Day Intervention for Residents
Brief Title: WILD 5 Wellness: A 30-Day Intervention for Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orange Park Medical Center (Other)
Responsible Party: Principal Investigator, AlexandraMary Kelada, DO, MPH, Internal medicine resident, Orange Park Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-014
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Resident Wellness; Burnout, Professional; Medical Residents; Mental Health Wellness 1; Mental Health Disorder; Resident Physician
MeSH Terms: conditions — Burnout, Professional; Mental Disorders | interventions — Health

STUDY DESIGN:
Intervention Model Description: WILD 5 Wellness is an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5-pronged wellness approach (Other): 30-day assessment of daily exercise, mindfulness, sleep, social connectedness, and nutrition
  Interventions: Behavioral: Wellness

INTERVENTIONS:
Behavioral: Wellness — Assess the feasibility of an integrated, prescriptive, and trackable wellness intervention amongst residents at Orange Park Medical Center (OPMC) by combining five wellness elements including: exercise, mindfulness, sleep, social connectedness, and nutrition.

SUMMARY:
The purpose of this study is to explore the efficacy and feasibility of an integrated, prescriptive, and trackable wellness intervention amongst resident physicians combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition.

DETAILED DESCRIPTION:
Data from the initial pilot of Wild 5 Wellness data reported at the Annual US Psychiatric Congress Meeting demonstrated positive results with their 30-day intervention: This study uses compelling proof that even a non-medication, self-directed, low cost 30-day intervention, focusing on mental wellness offers clinically significant help with mood, anxiety, mindfulness, sleep, social connectivity, and emotional eating (Jain et al., 2015)

The purpose of this study is to explore the efficacy and feasibility of an integrated, prescriptive, and trackable wellness intervention amongst residents at Orange Park Medical Center (OPMC) by combining five wellness elements including: exercise, mindfulness, sleep, social connectedness, and nutrition.

Data will be collected to evaluate participants' adherence and response to a 5-pronged 30-day wellness intervention. It is expected that this 30-day integrated, prescriptive, and trackable program will be found to be an efficacious wellness intervention among residents at OPMC.

To the best of our knowledge, even though there is abundant research supporting each of the WILD 5 Wellness elements (exercise, mindfulness, sleep, social connectedness, and nutrition) individually, there is no research exploring the effectiveness of an integrated, prescriptive, and trackable wellness intervention combining these five elements. Therefore, this work will be unique in that it will collect both objective and subjective data to assess the feasibility and effectiveness of this type of wellness intervention. It will lend support to the growing body of research on the efficacy of wellness interventions for a variety of different health conditions, as well as a residency-based population. Finally, it is hoped that positive results will yield increased access to and utilization of this type of intervention, thereby improving resident wellness.

ELIGIBILITY:
Inclusion Criteria:

* participants must be enrolled residents at Orange Park Medical Center (OPMC).

Exclusion Criteria:

* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in overall combined wellness score | 0 and 31 days
  Change in overall combined wellness score

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | 0 and 31 days
  A self-reported depression scale used to assess severity of depression.
Change in Generalized Anxiety Disorder-7 (GAD-7) | 0 and 31 days
  A self-reported questionnaire used to assess anxiety symptoms.
Change in World Health Organization-5 (WHO-5) | 0 and 31 days
  A brief scale that measures mental well- being.
Change in The Sleep Condition Indicator (SCI) | 0 and 31 days
  A brief scale that evaluates insomnia disorder.
Change in The Social Connectedness Scale (SCS) | 0 and 31 days
  A brief scale that assesses the degree to which respondents feel connected to others.
Change in Eating and Appraisal Due to Emotions and Stress (EADES) | 0 and 31 days
  A scale assessing how individuals cope with and appraise stress in relation to food and eating.
Change in The WILD 5 Wellness Scale (W5WS) | 0 and 31 days
  A brief scale designed specifically for this project to measure wellness.
The Post-Program Participant Questionnaire | 31 days
  A brief post study survey that captures participants' opinions about WILD 5 Wellness: 90-Day Intervention, and subjective ranking of their overall wellness.

CONTACTS AND LOCATIONS:
Overall Officials: AlexandraMary Kelada, DO, MPH, Principal Investigator — Orange Park Medical Center
Locations (1):
- Orange Park Medical Center, Orange Park, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.